CLINICAL TRIAL: NCT04933305
Title: Correlation Between Microstructure of Ingestive Behavior and Body Weight Loss in Patients After Roux-en-Y Gastric Bypass
Brief Title: Microstructure of Ingestive Behavior and Body Weight Loss After Roux-en-Y Gastric Bypass
Acronym: Drinkometer
Status: Completed | Type: Observational
Sponsor: Marco Bueter (Other)
Collaborators: Dr. Alan Spector, Florida State University, Department of Psychology (Unknown)
Responsible Party: Sponsor-Investigator, Marco Bueter, Assistant Professor, PhD, Head of Bariatric and Endocrine Surgery, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2017-00756
Record Dates: First submitted 2021-06-15; First posted 2021-06-21 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Obesity; Food Deprivation; Bariatric Surgery; Roux-en-y Gastric Bypass; Ingestive Microstructure; Ingestive Behavior; Drinkometer
MeSH Terms: conditions — Obesity; Feeding Behavior | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RYGB patients: Patients that already received RYGB one year prior commencement of their participation in the study
  Interventions: Procedure: Roux-en-Y Gastric Bypass

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass — Laparoscopic surgical procedure

SUMMARY:
Studies of appetitive behavior in humans after RYGB have produced ambiguous results. It therefore remains unclear whether there are fundamental shifts in the palatability of high-fat and sugary foods after RYGB or simply a decrease in the appetitive drive to ingest them. Moreover, learning processes may play a role as changes in diet selection progress with time in rats after RYGB. However, direct measures of an altered food selection in humans after RYGB are rare and both the durability of the phenomenon as well as the role of experience for changes in food selection remain elusive.

DETAILED DESCRIPTION:
Introduction Bariatric surgery (BS) is currently the most effective treatment of severe obesity. BS has a pleiotropic effect on the body, involving changes in basic metabolic rate, gut hormones and bile acid levels, intestinal nerve signaling and microbiota composition. Overall, patients report to eat less, to feel less hungry and they often change their food preferences. Initial insights on food intake and appetite can be provided by indirect measurements such as verbal report of energy intake, food diaries, and dietary recall questionnaires. However, indirect measurements are vulnerable to inaccuracy and, at best, only offer an estimate of the patients' real behavior. Such methodological limitations can be improved by complementing existing findings with direct measurements of eating and drinking. There are only very few studies to date that have applied direct measurements of ingestive behavior in BS patients. These studies focused mainly on macronutrient composition within a cafeteria diet and on some motivational aspects of appetitive behavior. This might be due to the fact that the assessment of the temporal organization of ingestive behavior within a meal in humans poses significant methodological and conceptual challenges to researchers and study design. The investigators have recently developed and validated a drinkometer for humans, which may have great utility in the investigation of the specific behavioral variables that underlie the altered appetite control in obesity, and also to specify neural effects of various medical or surgical weight-loss interventions.

The aim of this exploratory pilot study is to investigate a possible correlation between the microstructure of ingestive behavior and body weight loss in patients after Roux-en-Y gastric bypass with a follow-up of 5 years.

Methods Prospective observational study in patients that already received a RYGB. 50 patients will be recruited to consume a ready-to-drink, energy-dense oral nutritional supplement (product: Resource 2.0+fibre, Nestle, Vevey, Switzerland) in a food deprived state, until reaching satiety. The novel drinkometer will be used to measure ingestive microstructure and overall intake, and anthropometric parameters (weight, height) will be measured as well. Visual analogue scales will be used to assess self-reported hunger, thirst, fullness, liking, nausea, and pain. The participants will be asked to estimate their intake at the end of each session. The study visits will take place at each postoperative yearly control visit. Only for one subgroup of 30 patients, one year after surgery, one second study visit will be organised after an interval of two weeks from the first visit. In order to avoid sex-driven major differences in ingestive microstructure, only female participants will be included in the study.

Statistical analysis The drinkometer data will be processed and filtered by an in-house developed algorithm in Matlab 2017 software. Results will be analysed using descriptive statistics and statistical tests in RStudio software version 3.5.1.

Potential outcomes Any comprehensive understanding of how BS affects food intake requires a detailed analysis of the ingestive behavior itself, not simply the measurement of the outcome of the behavior. In other words, the information on how the food is consumed is equally or even more important than the information on how much food has been ingested. To the best of our knowledge, this is the first time that drinking microstructure in humans will be recorded and analyzed with a five-year follow-up in BS patients. Results will confirm if, in the long term, the microstructure of ingestive behavior might have a correlation with body weight loss or regain and hence be used as a predictor of surgery outcome. Further, this exploratory study may generate hypothesis on behavioral changes that occur following BS. Any treatment that affects total intake - e.g. BS - can be entirely viewed as function of its single components such as size and number of sucking bursts which then can provide relevant information e.g. on the motivational aspects of the ingestive behavior. The investigators expect to find at least two type of ingestive behaviours among study participants, one that would correlated with sustained body weight loss and one that would correlate with body weight regain.

Regardless of which outcomes are obtained, this innovative experiment will be a critical and a novel test of the explicit experience of humans with a high-sugar high-fat liquid meal after RYGB and its potential role for the understanding possible mechanisms determining postoperative outcomes, such as weight loss.

ELIGIBILITY:
Inclusion Criteria:

* received RYGB
* ability to provide inform consent

Exclusion Criteria:

* lactose intolerance
* diabetes
* immunosuppression
* pregnancy / lactation
* use of weight-loss medication
* history of previous visceral surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult females with severe obesity that underwent RYGB
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Correlation between microstructure of ingestive behavior and body weight loss | one year after surgery
  Pearson correlation coefficient for the linear relationship between microstrutural parameters of ingestive behavior and body weight loss one year after RYGB surgery

SECONDARY OUTCOMES:
Stability of the microstructure of ingestive behavior | fourteen days
  Significance of paired difference and equality tests for macrostructural parameters of ingestive behavior of the entire study population measured twice with an interval of fourteen days.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bueter, MD, DPhil, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gero D, File B, Justiz J, Steinert RE, Frick L, Spector AC, Bueter M. Drinking microstructure in humans: A proof of concept study of a novel drinkometer in healthy adults. Appetite. 2019 Feb 1;133:47-60. doi: 10.1016/j.appet.2018.08.012. Epub 2018 Sep 1. PMID 30179650
- [Background] Gero D, Steinert RE, le Roux CW, Bueter M. Do Food Preferences Change After Bariatric Surgery? Curr Atheroscler Rep. 2017 Sep;19(9):38. doi: 10.1007/s11883-017-0674-x. PMID 28779431
- [Background] Mathes CM, Bohnenkamp RA, Blonde GD, Letourneau C, Corteville C, Bueter M, Lutz TA, le Roux CW, Spector AC. Gastric bypass in rats does not decrease appetitive behavior towards sweet or fatty fluids despite blunting preferential intake of sugar and fat. Physiol Behav. 2015 Apr 1;142:179-88. doi: 10.1016/j.physbeh.2015.02.004. Epub 2015 Feb 3. PMID 25660341
- [Background] Spector AC, Klumpp PA, Kaplan JM. Analytical issues in the evaluation of food deprivation and sucrose concentration effects on the microstructure of licking behavior in the rat. Behav Neurosci. 1998 Jun;112(3):678-94. doi: 10.1037//0735-7044.112.3.678. PMID 9676983
- [Background] Johnson AW. Characterizing ingestive behavior through licking microstructure: Underlying neurobiology and its use in the study of obesity in animal models. Int J Dev Neurosci. 2018 Feb;64:38-47. doi: 10.1016/j.ijdevneu.2017.06.012. Epub 2017 Jul 3. PMID 28684308